CLINICAL TRIAL: NCT01713946
Title: A Three-arm, Randomized, Double-blind, Placebo-controlled Study of the Efficacy and Safety of Two Trough-ranges of Everolimus as Adjunctive Therapy in Patients With Tuberous Sclerosis Complex (TSC) Who Have Refractory Partial-onset Seizures
Brief Title: A Placebo-controlled Study of Efficacy & Safety of 2 Trough-ranges of Everolimus as Adjunctive Therapy in Patients With Tuberous Sclerosis Complex (TSC) & Refractory Partial-onset Seizures
Acronym: EXIST-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRAD001M2304; 2011-000860-90 (EudraCT Number)
Record Dates: First submitted 2012-10-09; First posted 2012-10-25 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Tuberous Sclerosis Complex-associated Refractory Seizures
Keywords: TSC seizures; TSC epilepsy; mTOR inhibitor; RAD001; Everolimus
MeSH Terms: interventions — Everolimus; Anticonvulsants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Everolimus LT target of 3 - 7 ng/mL (Experimental): Participants received everolimus dispersible tablets for oral suspension with titration to a low trough (LT) range of 3 to 7 ng/mL plus 1 to 3 antiepileptic drugs.
  Interventions: Drug: RAD001; Drug: Antiepileptic drug (1 to 3 only); Drug: open label RAD001 (only used for post-extension phase)
- Everolimus HT target of 9 -15 ng/mL (Experimental): Participants received everolimus dispersible tablets for oral suspension with titration to a high trough (HT) range of 9 to 15 ng/mL plus 1 to 3 antiepileptic drugs.
  Interventions: Drug: RAD001; Drug: Antiepileptic drug (1 to 3 only); Drug: open label RAD001 (only used for post-extension phase)
- Placebo (Placebo Comparator): Participants received placebo plus 1 to 3 antiepileptic drugs.
  Interventions: Drug: Placebo; Drug: Antiepileptic drug (1 to 3 only); Drug: open label RAD001 (only used for post-extension phase)

INTERVENTIONS:
Drug: RAD001 — Everolimus tablets for oral suspension (dispersible tablets) were packaged as 2 mg tablets in blister packs and placed in boxes with color-coded labels, color 1 or color 2.
  Other Names: everolimus
  Arms: Everolimus HT target of 9 -15 ng/mL; Everolimus LT target of 3 - 7 ng/mL
Drug: Placebo — Placebo tablets for oral suspension (dispersible tablets) were packaged as 2 mg tablets in blister packs and placed in boxes with color-coded labels, color 1 or color 2.
  Arms: Placebo
Drug: Antiepileptic drug (1 to 3 only) — no more than any 3 of the listed antiepileptic drugs could be taken with the study drug or placebo. List of allowed antiepileptic drugs were: valporic acid, carbamazepine, clobazam, N-desmethylclobazam, topiramate,TRI477, TRI476, clonazepam, zonisamide, phenobarbital, phenytoin
Drug: open label RAD001 (only used for post-extension phase) — everolimus tablets for oral suspension (dispersible tablets) were packaged as 2 mg tablets in blister backs in boxes with open label design and were taken during the Post-Extension phase, where all the participants, including those who were previously on placebo, took the 2mg tablets.
  Other Names: open label everolimus

SUMMARY:
This study evaluated the efficacy and safety of two trough-ranges of everolimus given as adjunctive therapy in patients with tuberous sclerosis complex (TSC) who had refractory partial-onset seizures.

The study consisted of 4 phases for each patient Baseline phase:[From Screening Week -8 (V1) to randomization visit at Week 0 (V2)], Core phase [from randomization at Week 0 (V2) to Week 18 (V11)], Extension phase [from Week 18 (V11) until 48 weeks after the last patient had completed the core phase] and Post Extension phase [from end of Extension phase to end of study].

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female between the ages of 2 and 65 years (except in Europe where minimum age will be 1).

  2. Clinically definite diagnosis of TSC per modified Gomez criteria 3. Diagnosis of partial-onset epilepsy according to the classification of the International League Against Epilepsy (1989) and revised in 2009.

  4. Uncontrolled partial-onset seizures; must meet the following:
  1. At least 16 reported quantifiable partial-onset seizures over the Baseline period with no continuous 21-day seizure-free period between Visit 1 (Screening Visit) and Visit 2 (Randomization visit), as per data captured in daily seizure diaries.
  2. Prior history of failure to control partial-onset seizures despite having been treated with two or more sequential regimens of single or combined antiepileptic drugs.
  3. Prior or concurrent use of vagal nerve stimulator (VNS) is allowed. If the patient is using VNS, device stimulator parameters must remain constant throughout the study.
  4. Prior epilepsy surgery is allowed if performed at least 12 months before study entry.

     5. Must be receiving one, two, or three AEDs at a stable dose for at least 4 weeks at the start of the 8-week prospective Baseline phase, remain on the same regimen throughout the Baseline phase, and intend to continue the same regimen throughout the 18-week double blind Core phase (rescue medications are permitted).

     6. If female of child bearing potential, documentation of negative pregnancy test at time of informed consent and must use highly effective contraception during the study and for 8 weeks after stopping treatment 7. Sexually active males must use a condom during intercourse while taking study drug, and for 8 weeks after stopping study treatment 8. Hepatic, renal and blood laboratory values within the following range at screening :

  <!-- -->

  1. AST and ALT levels < 2.5 x ULN
  2. serum bilirubin <1.5 × ULN (this limit does not apply to patients with an elevated indirect bilirubin, if they have Gilbert's Syndrome),
  3. serum creatinine < 1.5 x ULN
  4. hemoglobin ≥ 9 g/dL
  5. platelets ≥ 80,000/mm3
  6. absolute neutrophil count ≥ 1,000/mm3 9. Written informed consent. Subjects or their legal guardians must have the ability to comprehend the informed consent form and be willing to provide informed consent.

     10. Patient or caregiver must be able to reliably record seizures and keep a daily diary and recall adverse events.

     Exclusion Criteria:
* 1. Patients with seizures secondary to metabolic, toxic, infectious or psychogenic disorder or drug abuse or current seizures related to an acute medical illness.

  2. Presence of only non-motor partial seizures (NOT APPLICABLE per Amendment 2) 3. Patients with TSC who have SEGA in need of immediate surgical intervention. 4. Patients under 2 years of age with untreated infantile spasms. 5. Within 52 weeks prior to study entry, an episode of status epilepticus as defined in the protocol.

  6. Patients with history of seizure clusters (where individual seizures cannot be accurately counted according to the judgment of the investigator) occurring within 26 weeks prior to study entry.

  7. Patients who require rescue medication during the baseline phase for more than 6 days 8. Patients with non-TSC related progressive encephalopathy. 9. Patients who weigh less than 12 kg. 10. Patients with coexisting malignancies within the 3 years prior to randomization, except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.

  11. Patients with any severe and/or uncontrolled medical conditions at randomization such as:
  1. Symptomatic congestive heart failure of New York Heart Association Class III or IV, history of left ventricular ejection fraction (LVEF) < 50%, QTc interval >460ms, congenital QT syndrome, unstable angina pectoris, myocardial infarction within 6 months of study entry, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease.
  2. Significant symptomatic deterioration of lung function
  3. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, malabsorption syndrome or small bowel resection).
  4. liver disease such as cirrhosis, decompensated liver disease, and chronic hepatitis
  5. Uncontrolled diabetes as defined by fasting serum glucose > 1.5 × ULN.
  6. Active skin, mucosa, ocular or GI disorders of Grade > 1.
  7. Active (acute or chronic) or uncontrolled severe infections.
  8. A known history of HIV seropositivity or other active viral infections. 12. Patients with an active, bleeding diathesis. 13. Patient with uncontrolled hyperlipidemia: fasting serum cholesterol > 300 mg/dL OR >7.75 mmol/L AND fasting triglycerides > 2.5 x ULN.

     14. Patients who have had a major surgery or significant traumatic injury within 4 weeks of study entry.

     15. Patients with a prior history of organ transplant. 16. Patients receiving more than 3 antiepileptic drugs at any time in the baseline phase or at randomization or who change the dose of the AEDs during 4 weeks before screening or during the baseline period.

     17. Patients being treated with felbamate, unless treatment has been continuous for ≥ 1 year.

     18. Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of study entry (including chemotherapy, radiation therapy, antibody based therapy, etc.).

     19. Prior treatment with any investigational drug within the preceding 4 weeks prior to study entry.

     20. Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent at study entry. Topical or inhaled corticosteroids are allowed.

     21. Patients who have received prior treatment with a systemic mTOR inhibitor (sirolimus, temsirolimus, everolimus) within 24 months of study entry. Patients who have received prior treatment with a topical mTOR inhibitor (sirolimus, temsirolimus, everolimus) within 4 weeks of study entry.

     22. Patients with a known hypersensitivity to everolimus or other rapamycin-analogues (sirolimus, temsirolimus) or to its excipients.

     23. Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study 24. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.

     25. Patients with a Score of 4 or 5 on the Suicidal Ideation item within 2 years of Screening, or any "yes" on the Suicidal Behavior item of the Columbia-Suicide Severity Rating Scale at Screening or Baseline , who upon follow up with a healthcare professional are found to be severely depressed or suicidal.

     26. Maintenance of a diet consisting of <40 g of carbohydrate per day within 3 months of screening

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2013-04-29 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (96):
- United States (22):
  - University of Alabama at Birmingham SC, Birmingham, Alabama
  - TGen/APNNA, Phoenix, Arizona
  - University of California at Los Angeles SC, Los Angeles, California
  - Children's Hospital Oakland SC, Oakland, California
  - Children's Hospital of Orange County SC, Orange, California
  - Rady Children's Hospital SC, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Childrens Medical Center SC, Hartford, Connecticut
  - University of Chicago SC - 2, Chicago, Illinois
  - Kennedy Krieger Institute SC, Baltimore, Maryland
  - Children's Hospital Boston SC, Boston, Massachusetts
  - Minnesota Epilepsy Group - PA SC, Saint Paul, Minnesota
  - Washington University School of Medicine SC-2, St Louis, Missouri
  - Morristown Memorial Hospital SC-2, Morristown, New Jersey
  - New York University Medical Center SC-3, New York, New York
  - Cincinnati Children's Hospital Medical Center SC, Cincinnati, Ohio
  - Oregon Health and Science University SC - 3, Portland, Oregon
  - Children's Hospital of Philadelphia SC, Philadelphia, Pennsylvania
  - LeBonheur Childrens Medical Group SC, Memphis, Tennessee
  - Texas Scottish Rite Hospital for Children Texas Scottish, Dallas, Texas
  - Texas Children s Hospital SC, Houston, Texas
  - The University of Texas Medical School-Houston SC, Houston, Texas
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Córdoba
- Australia (3):
  - Novartis Investigative Site, Randwick, New South Wales
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Perth, Western Australia
- Belgium (4):
  - Novartis Investigative Site, Jette, Brussels Capital
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Canada (2):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Montreal, Quebec
- Colombia (3):
  - Novartis Investigative Site, Cali, Valle del Cauca Department
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Medellín
- Novartis Investigative Site, Aarhus, Denmark
- France (6):
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Strasbourg
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Kehl-Kork
  - Novartis Investigative Site, Kiel
- Greece (2):
  - Novartis Investigative Site, Ioannina, GR
  - Novartis Investigative Site, Athens
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Nyíregyháza
- Novartis Investigative Site, Dublin, Ireland
- Italy (8):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
- Japan (6):
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Izumi, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Shizuoka, Shizuoka
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Osaka
- Novartis Investigative Site, Guadalajara, Jalisco, Mexico
- Netherlands (3):
  - Novartis Investigative Site, Heeze
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Utrecht
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Warsaw, Poland
- Russia (3):
  - Novartis Investigative Site, Samara, Samara Oblast
  - Novartis Investigative Site, Voronezh, Voronezh Oblast
  - Novartis Investigative Site, Moscow
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Taiwan (3):
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
- United Kingdom (7):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Buckinghamshire
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Sheffield
  - Novartis Investigative Site, York

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Curatolo P, Franz DN, Lawson JA, Yapici Z, Ikeda H, Polster T, Nabbout R, de Vries PJ, Dlugos DJ, Fan J, Ridolfi A, Pelov D, Voi M, French JA. Adjunctive everolimus for children and adolescents with treatment-refractory seizures associated with tuberous sclerosis complex: post-hoc analysis of the phase 3 EXIST-3 trial. Lancet Child Adolesc Health. 2018 Jul;2(7):495-504. doi: 10.1016/S2352-4642(18)30099-3. Epub 2018 May 24. PMID 30169322
- [Derived] French JA, Lawson JA, Yapici Z, Ikeda H, Polster T, Nabbout R, Curatolo P, de Vries PJ, Dlugos DJ, Berkowitz N, Voi M, Peyrard S, Pelov D, Franz DN. Adjunctive everolimus therapy for treatment-resistant focal-onset seizures associated with tuberous sclerosis (EXIST-3): a phase 3, randomised, double-blind, placebo-controlled study. Lancet. 2016 Oct 29;388(10056):2153-2163. doi: 10.1016/S0140-6736(16)31419-2. Epub 2016 Sep 6. PMID 27613521
- [Derived] Goyer I, Dahdah N, Major P. Use of mTOR inhibitor everolimus in three neonates for treatment of tumors associated with tuberous sclerosis complex. Pediatr Neurol. 2015 Apr;52(4):450-3. doi: 10.1016/j.pediatrneurol.2015.01.004. Epub 2015 Jan 14. PMID 25682485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 355 patients were planned to be enrolled and a total of 366 patients were randomized: 117 to the everolimus targeted low-trough arm (LT), 130 to the everolimus targeted high-trough (HT) arm, and 119 to treatment with placebo.
Groups:
- Everolimus LT Target of 3 to 7 ng/mL: Participants were randomized to receive everolimus dispersible tablets for oral suspension with titration to a low trough (LT) range of 3 to 7 ng/mL
- Everolimus HT Target of 9 to 15 ng/mL: Participants were randomized to receive everolimus dispersible tablets for oral suspension with titration to a high trough (HT) range of 9 to 15 ng/mL
- Placebo: Participants who received placebo dispersible tablets for oral suspension at study start and switched to everolimus in Extension.
Period: Overall Study
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo
Started | 117 | 130 | 119 (Of the 119 patients initially randomized to the Placebo arm, 5 patients never switched to everolimus)
Completed Core Phase | 110 | 122 | 114
Continued in Ext. Phase | 110 | 119 | 114
Completed Ext. Phase | 79 | 92 | 81
Continued in Post-Ext. Phase | 78 | 90 | 81
Completed Post-Ext Phase | 74 | 85 | 75
Did Not Continue in Ext Phase | 0 | 3 | 0
Did Not Cont. in Post-Ext Phase | 1 | 2 | 0
Completed | 74 | 85 | 75
Not Completed | 43 | 45 | 44
Not completed — Death | 0 | 2 | 2
Not completed — Adverse Event | 19 | 14 | 13
Not completed — Withdrawal by Subject | 12 | 12 | 8
Not completed — Lack of Efficacy | 8 | 8 | 14
Not completed — Protocol Violation | 2 | 4 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Administrative problems | 1 | 0 | 0
Not completed — Did not continue in Ext | 0 | 3 | 0
Not completed — Did not continue in Post-Ext. Phase | 1 | 2 | 0
Not completed — Patients never switched to everolimus | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Groups:
- Placebo: Participants were randomized to receive placebo dispersible tablets for oral suspension.
- Total: Total of all reporting groups
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo | Total
Number analyzed (Participants) | 117 | 130 | 119 | 366
Age, Continuous [Median (Full Range); unit: years] — Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
  years | 9.72 [2.2 to 56.3] | 10.08 [2.3 to 50.5] | 10.34 [2.2 to 52.0] | 10.06 [2.2 to 56.3]
Age, Customized [Count of Participants; unit: Participants] — Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
  Participants
    < 6 years | 33 | 37 | 34 | 104
    6 to <12 years | 37 | 39 | 37 | 113
    12 to <18 years | 26 | 31 | 25 | 82
    18 to <65 years | 21 | 23 | 23 | 67
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
  Participants
    Female | 53 | 65 | 58 | 176
    Male | 64 | 65 | 61 | 190
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
  Participants
    Caucasian | 76 | 84 | 77 | 237
    Asian | 29 | 31 | 27 | 87
    Black | 2 | 1 | 1 | 4
    Native American | 0 | 1 | 0 | 1
    Pacific Islander | 1 | 0 | 0 | 1
    Other | 9 | 13 | 14 | 36
Weight [Mean (Standard Deviation); unit: kg] — Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
  kg | 38.69 (22.802) | 40.75 (27.267) | 40.50 (24.923) | 40.01 (25.093)
Height [Mean (Standard Deviation); unit: cm] — Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
  cm | 135.65 (26.171) | 136.25 (28.234) | 135.67 (27.097) | 135.87 (27.145)
Body surface area [Mean (Standard Deviation); unit: m^2] — Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
  m^2 | 1.18 (0.437) | 1.20 (0.501) | 1.20 (0.476) | 1.20 (0.472)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
  kg/m^2 | 19.29 (5.283) | 19.56 (6.233) | 19.78 (5.484) | 19.55 (5.689)

OUTCOME MEASURES:

1. Primary Outcome: Core Phase: European Medicine Agency (EMA): Seizure Frequency Response Rate
Description: Comparison of response rates in the everolimus low-trough treatment arm (3-7 ng/mL), high-trough treatment arm (9-15 ng/mL) and placebo arm. Response means at least a 50% reduction from baseline in partial-onset seizure frequency during the maintenance period of the core phase.
Time Frame: Baseline (8-week period before randomization), Week 7 to 18 (12-week maintenance period of the core phase)
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo
Number analyzed (Participants) | 117 | 130 | 119
Percentage of responders | 28.2 [20.3 to 37.3] | 40.0 [31.5 to 49.0] | 15.1 [9.2 to 22.8]
Statistical Analysis 1: Comparison: Everolimus LT Target of 3 to 7 ng/mL vs Placebo; Test type: Superiority; p = 0.008, Bonferroni-Holm; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.16 to 4.20]
Statistical Analysis 2: Comparison: Everolimus HT Target of 9 to 15 ng/mL vs Placebo; Test type: Superiority; p < 0.001, Bonferroni-Holm; Odds Ratio (OR) = 3.93, 95% CI 2-sided [2.10 to 7.32]

2. Primary Outcome: Core Phase: Food & Drug Administration (FDA): Percentage Change From Baseline in Partial Onset-seizure Frequency
Description: Comparison of median percent change from baseline in weekly seizure frequency in the everolimus low-trough treatment arm (3-7 ng/mL), high-trough treatment arm (9-15 ng/mL) and placebo arm during maintenance period of the core phase. Percentage change from baseline in average weekly seizure frequency during the maintenance period of the Core phase (SFcfb) = 100 × (SFB - SFM) ÷ SFB where:
  SFB is the average weekly seizure frequency in the Baseline phase SFM is the average weekly seizure frequency in the maintenance period of the Core phase A positive percentage change from baseline (SFcfb) means a reduction in seizure frequency whereas a negative percentage change from baseline (SFcfb) means an increase in seizure frequency.
Time Frame: Baseline (8-week period before randomization), Week 7 to 18 (12-week maintenance period of the core phase)
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization
Measure: Median (95% Confidence Interval); unit: Percentage change from baseline
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo
Number analyzed (Participants) | 117 | 130 | 119
Percentage change from baseline | 29.29 [18.82 to 41.88] | 39.55 [35.03 to 48.74] | 14.86 [0.11 to 21.71]
Statistical Analysis 1: Comparison: Everolimus LT Target of 3 to 7 ng/mL vs Placebo; Test type: Superiority; p = 0.003, Bonferroni-Holm; Median Difference (Final Values) = 15.96, 95% CI 2-sided [1.98 to 31.68]
Statistical Analysis 2: Comparison: Everolimus HT Target of 9 to 15 ng/mL vs Placebo; Test type: Superiority; p < 0.001, Bonferroni-Holm; Odds Ratio (OR) = 27.46, 95% CI 2-sided [16.36 to 43.36]

3. Secondary Outcome: Percentage of Seizure-free Patients During the Maintenance Period of the Core Phase
Description: Comparison of seizure freedom (100% reduction in seizure frequency) in the everolimus low-trough treatment arm (3-7 ng/mL), high-trough treatment arm (9-15 ng/mL) and placebo arm during maintenance period of the core phase. Seizure free means a 100% reduction from baseline in partial-onset seizure frequency during maintenance period of the core phase.
Time Frame: Baseline (8-week period before randomization), Week 7 to 18 (12-week maintenance period of the core phase)
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization
Measure: Number (95% Confidence Interval); unit: Percentage of seizure-free participants
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo
Number analyzed (Participants) | 117 | 130 | 119
Percentage of seizure-free participants | 5.1 [1.9 to 10.8] | 3.8 [1.3 to 8.7] | 0.8 [0.0 to 4.6]
Statistical Analysis 1: Comparison: Everolimus LT Target of 3 to 7 ng/mL vs Placebo; Test type: Superiority; Odds Ratio (OR) = 6.55, 95% CI 2-sided [0.77 to 55.73]
Statistical Analysis 2: Comparison: Everolimus HT Target of 9 to 15 ng/mL vs Placebo; Test type: Superiority; Odds Ratio (OR) = 4.99, 95% CI 2-sided [0.57 to 44.03]

4. Secondary Outcome: Core Phase: Percentage of Patients With at Least a 25% Reduction in Seizure Frequency
Description: Comparison of percentage of patients with at least ≥ 25% reduction in seizure frequency in the everolimus low-trough treatment arm (3-7 ng/mL), high-trough treatment arm (9-15 ng/mL) and placebo arm during maintenance period of the core phase. At least 25% reduction from baseline in partial-onset seizure frequency during maintenance period of the core phase.
Time Frame: Baseline (8-week period before randomization), Week 7 to 18 (12-week maintenance period of the core phase)
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo
Number analyzed (Participants) | 117 | 130 | 119
Percentage of participants | 52.1 [42.7 to 61.5] | 70.0 [61.3 to 77.7] | 37.8 [29.1 to 47.2]
Statistical Analysis 1: Comparison: Everolimus LT Target of 3 to 7 ng/mL vs Placebo; Test type: Superiority; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.05 to 2.97]
Statistical Analysis 2: Comparison: Everolimus HT Target of 9 to 15 ng/mL vs Placebo; Test type: Superiority; Odds Ratio (OR) = 3.82, 95% CI 2-sided [2.25 to 6.48]

5. Secondary Outcome: Core Phase: Distribution of Reduction From Baseline in Seizure Frequency
Description: Comparison of percentage of patients in six categories of seizure reduction from baseline (≤ -25% (exacerbation); > -25% to < 25% (no change); ≥ 25% to < 50%; ≥ 50% to < 75%; ≥ 75% to < 100%; 100% (seizure-freedom)) in the everolimus low-trough treatment arm (3-7 ng/mL), high-trough treatment arm (9-15 ng/mL) and placebo arm during maintenance period of the core phase
Time Frame: Baseline (8-week period before randomization), Week 7 to 18 (12-week maintenance period of the core phase)
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo
Number analyzed (Participants) | 117 | 130 | 119
Percentage of participants
  100% (seizure free) | 5.1 | 3.8 | 0.8
  ≥ 75 to <100 (75% responder) | 6.0 | 15.4 | 5.0
  ≥ 50 to <75 (50% responder) | 17.1 | 20.8 | 9.2
  ≥ 25 to <50 (25% responder) | 23.9 | 30.0 | 22.7
  >-25 to <25 (No change) | 35.0 | 18.5 | 41.2
  ≤ -25 (Exacerbation) | 12.8 | 11.5 | 20.2
  Missing (missing) | 0.0 | 0.0 | 0.8

6. Secondary Outcome: Core Phase: Changes From Baseline in Number of Seizure-free Days
Description: Comparison of seizure-free days relative to baseline in the everolimus low-trough treatment arm (3-7 ng/mL), high-trough treatment arm (9-15 ng/mL) and placebo arm during maintenance period of the core phase
Time Frame: Baseline (8-week period before randomization), Week 7 to 18 (12-week maintenance period of the core phase)
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization
Measure: Median (Full Range); unit: Number of seizure-free days -per 28 days
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo
Number analyzed (Participants) | 117 | 130 | 119
Number of seizure-free days -per 28 days | 2.00 [-23.1 to 27.7] | 4.01 [-10.0 to 27.5] | 0.47 [-13.4 to 21.8]
Statistical Analysis 1: Comparison: Everolimus LT Target of 3 to 7 ng/mL vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-0.4 to 3.1]
Statistical Analysis 2: Comparison: Everolimus HT Target of 9 to 15 ng/mL vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 4.2, 95% CI 2-sided [2.5 to 5.9]

7. Secondary Outcome: Core Phase: Probability That a Patient Remains On-treatment up to a Specified Time Point
Description: Comparison of time to treatment discontinuation in the everolimus low-trough treatment arm (3-7 ng/mL), high-trough treatment arm (9-15 ng/mL) and placebo arm during the core phase. Treatment duration is defined as the time from randomization until the date of permanent study treatment discontinuation (for any reason) at any time during the Core phase.
  The percentage event-free probability estimate is the estimated probability that a patient will remain on-treatment up to a specified time point (Week 6, 12, 18)
Time Frame: Week 6, Week 12, Week 18
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization
Measure: Number (95% Confidence Interval); unit: Percentage event-free prob. estimates
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo
Number analyzed (Participants) | 117 | 130 | 119
Percentage event-free prob. estimates
  Week 6 | 97.4 [92.3 to 99.2] | 96.2 [91.0 to 98.4] | 99.2 [94.2 to 99.9]
  Week 12 | 95.7 [90.0 to 98.2] | 95.4 [90.0 to 97.9] | 97.5 [92.4 to 99.2]
  Week 18 | 70.1 [60.9 to 77.5] | 71.5 [62.9 to 78.5] | 75.6 [66.9 to 82.4]
Statistical Analysis 1: Comparison: Everolimus LT Target of 3 to 7 ng/mL vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.27, 95% CI 2-sided [0.77 to 2.07]
Statistical Analysis 2: Comparison: Everolimus HT Target of 9 to 15 ng/mL vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.74 to 1.96]

8. Secondary Outcome: Core Phase: Change From Baseline in the QOLCE Overall Quality-of-life Score for Patients <11 Years
Description: Comparison of quality of life in the everolimus (from 3 age specific questionnaires) low-trough treatment arm (3-7 ng/mL), high-trough treatment arm (9-15 ng/mL) and placebo arm at the end of the core phase. The Quality of Life Childhood Epilepsy (QOLCE) questionnaire, used for patients < 11 years at baseline, was completed by the patient's parent or caregiver. It consists of 16 subscales (13 multi-item scales and 3 single item scales) and one overall quality-of-life score. Scores range from 0-100, with higher scores corresponding to improved QoL. The Overall Quality of Life Score is computed by adding each subscale score for each individual and then dividing by 16.
Time Frame: Baseline, Week 18
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo
Number analyzed (Participants) | 65 | 69 | 63
scores on a scale
  Baseline: number analyzed (Participants) | 63 | 68 | 55
  Baseline | 52.3 [26 to 75] | 56.5 [26 to 76] | 55.3 [33 to 74]
  End of Core Phase: number analyzed (Participants) | 56 | 56 | 50
  End of Core Phase | 53.6 [24 to 79] | 59.5 [36 to 78] | 57.2 [20 to 77]
  Change from Baseline: number analyzed (Participants) | 55 | 56 | 47
  Change from Baseline | 0.2 [-25 to 24] | 0.0 [-19 to 18] | 1.0 [-18 to 28]
Statistical Analysis 1: Comparison: Everolimus LT Target of 3 to 7 ng/mL vs Placebo; Test type: Superiority; Difference in least square means = -1.1, 95% CI 2-sided [-4.4 to 2.1]
Statistical Analysis 2: Comparison: Everolimus HT Target of 9 to 15 ng/mL vs Placebo; Test type: Superiority; Difference in least square means = 1.0, 95% CI 2-sided [-2.2 to 4.3]

9. Secondary Outcome: Core Phase: Change From Baseline in the QOLIE-AD-48 Overall Quality-of-life Score for Patients >=11 to 18 Years
Description: Comparison of quality of life (from 3 age specific questionnaires) in the everolimus low-trough treatment arm (3-7 ng/mL), hightrough treatment arm (9-15 ng/mL) and placebo arm at the end of the core phase. The Quality of Life in Epilepsy Inventory for Adolescents-48 (QOLIE-AD-48) is a survey of health-related quality of life for adolescents 11 to 18 years of age with epilepsy. The QOLIE-AD-48 is completed by the patient. It contains 48 items which assess 8 subscales. Scores range from 0-100, with higher scores corresponding to improved QoL. The overall quality of life score is obtained by summing a linear combination of the 8 subscale scores, where each subscale is multiplied by a relative weight that is provided in the original publication.
Time Frame: Baseline, Week 18
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo
Number analyzed (Participants) | 31 | 38 | 33
scores on a scale
  Baseline: number analyzed (Participants) | 13 | 15 | 14
  Baseline | 56.1 [43 to 86] | 58.8 [35 to 81] | 59.6 [13 to 88]
  End of Core Phase: number analyzed (Participants) | 13 | 13 | 12
  End of Core Phase | 58.5 [47 to 89] | 60.7 [46 to 74] | 65.4 [29 to 87]
  Change from Baseline: number analyzed (Participants) | 12 | 13 | 12
  Change from Baseline | 4.7 [-11 to 11] | 5.8 [-13 to 38] | 7.2 [-18 to 25]
Statistical Analysis 1: Comparison: Everolimus LT Target of 3 to 7 ng/mL vs Placebo; Test type: Superiority; Difference in least square means = -2.1, 95% CI 2-sided [-10.5 to 6.2]
Statistical Analysis 2: Comparison: Everolimus HT Target of 9 to 15 ng/mL vs Placebo; Test type: Superiority; Difference in least square means = 0.4, 95% CI 2-sided [-7.8 to 8.6]

10. Secondary Outcome: Core Phase: Change From Baseline in the QOLIE-31-P Overall Quality-of-life Score for Patients Aged >=18 Years
Description: Comparison of quality of life (from 3 age specific questionnaires) in the everolimus low-trough treatment arm (3-7 ng/mL), hightrough treatment arm (9-15 ng/mL) and placebo arm at the end of the core phase. The Quality of Life in Epilepsy Inventory-31-Problems (QOLIE-31-P) is a survey of health-related quality of life for adults with epilepsy. The QOLIE-31-P is completed by the patient. It contains 39 items, of which a total of 30 are used to make up 7 different subscales. Scores range from 0-100, with higher scores indicating a greater level of functioning and QoL. The overall quality of life score is obtained by summing a linear combination of the 7 subscale scores, where each subscale is multiplied by a relative weight that is obtained from the patient's answer to 7 items of this questionnaire.
Time Frame: Baseline, Week 18
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo
Number analyzed (Participants) | 21 | 23 | 23
scores on a scale
  Baseline: number analyzed (Participants) | 11 | 11 | 15
  Baseline | 39.5 [13 to 64] | 43.2 [5 to 89] | 43.6 [11 to 83]
  End of Core Phase: number analyzed (Participants) | 10 | 11 | 12
  End of Core Phase | 48.6 [11 to 54] | 37.1 [6 to 97] | 54.8 [26 to 90]
  Change from Baseline: number analyzed (Participants) | 10 | 11 | 12
  Change from Baseline | -0.5 [-17 to 34] | 0.4 [-47 to 20] | 5.3 [-16 to 36]
Statistical Analysis 1: Comparison: Everolimus LT Target of 3 to 7 ng/mL vs Placebo; Test type: Superiority; Difference in least square means = -2.8, 95% CI 2-sided [-17.9 to 12.3]
Statistical Analysis 2: Comparison: Everolimus HT Target of 9 to 15 ng/mL vs Placebo; Test type: Superiority; Difference in least square means = -7.7, 95% CI 2-sided [-22.0 to 6.6]

11. Secondary Outcome: Core Phase: Change From Baseline in the Overall Vineland-II Adaptive Behavior Composite (ABC) Score
Description: Comparison of adaptive functioning using the VABS-II composite score in the everolimus low-trough treatment arm (3-7 ng/mL), high-trough treatment arm (9-15 ng/mL) and placebo arm. The Vineland II assesses an individual's development of personal independence & social responsibility. The questionnaire contains 433 items which assess 15 subdomains organized into the five domains of Communication, Daily Living Skills, Socialization, Motor Skills and Maladaptive Behavior. The overall Adaptive Behavior Composite (ABC) score is obtained by summing the standard scores of the first four domain scores for patients aged less than 7 years, or the first 3 domain scores for patients aged 7 or older (the Maladaptive Behavior domain is optional). The ABC standard score ranges from 20 to 160 with a mean of 100 and a standard deviation of 15. Higher scores correspond to improved adaptive level. Note that 2 questionnaires with ABC scores<20 (data issues) were included in this analysis.
Time Frame: Baseline, 18 weeks
Population: The safety Set comprised all patients who received at least one dose of study treatment and had at least one post-baseline safety assessment in the Core phase (where the statement that a patient had no AE constitutes a safety assessment).
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo
Number analyzed (Participants) | 75 | 93 | 76
scores on a scale
  Baseline: number analyzed (Participants) | 34 | 34 | 32
  Baseline | 58.00 [20.0 to 112.0] | 56.50 [20.0 to 102.0] | 55.00 [20.0 to 103.0]
  End of Core Phase: number analyzed (Participants) | 28 | 39 | 31
  End of Core Phase | 54.00 [6.0 to 121.0] | 55.00 [20.0 to 111.0] | 55.00 [20.0 to 105.0]
  Change from Baseline: number analyzed (Participants) | 18 | 23 | 23
  Change from Baseline | -1.00 [-21.0 to 15.0] | 0.00 [-13.0 to 15.0] | 0.00 [-12.0 to 10.0]

12. Secondary Outcome: Long Term Evaluation: Effect of Everolimus Over Time in the Overall Vineland-II Adaptive Behavior Composite (ABC) Score
Description: as for outcome 11
Time Frame: Baseline, Weeks 18, 42, 66 and 90
Population: The Long Term Evaluation (LTE) efficacy set consists of all patients who received at least one dose of everolimus and had at least one efficacy assessment while on everolimus.
Measure: Median (Full Range); unit: scores on a scale
Groups:
- Everolimus Long Term Evaluation (LTE): Participants who were treated with everolimus either in the Core or Extension phases of the study and were evaluated for longer term safety and efficacy.
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo | Everolimus Long Term Evaluation (LTE)
Number analyzed (Participants) | 0 | 0 | 0 | 239
scores on a scale
  Baseline: number analyzed (Participants) | 0 | 0 | 0 | 88
  Baseline |  |  |  | 56.00 [20.0 to 112.0]
  Week 18: number analyzed (Participants) | 0 | 0 | 0 | 94
  Week 18 |  |  |  | 53.50 [4.0 to 121.0]
  Week 42: number analyzed (Participants) | 0 | 0 | 0 | 94
  Week 42 |  |  |  | 55.50 [20.0 to 111.0]
  Week 66: number analyzed (Participants) | 0 | 0 | 0 | 88
  Week 66 |  |  |  | 57.00 [20.0 to 112.0]
  Week 90: number analyzed (Participants) | 0 | 0 | 0 | 66
  Week 90 |  |  |  | 49.50 [20.0 to 150.0]

13. Secondary Outcome: Core Phase: Change From Baseline in Wechsler Nonverbal Composite Score
Description: The brief version of the WNV consists of a 2-subtest battery: only Matrices and Recognition subtests for patients under 8, and Matrices and Spatial Span subtests for patients aged 8 to 21. Based on the raw scores obtained from the subtests, standardized z-scores were calculated for each subtest using the following formula: Zscore = (X - b)/Sb where X is the raw score of the subtest, b and Sb represent the mean and standard deviation respectively of the subtest score recorded at baseline for the study population. The composite WNV score was computed by summing up the Z-scores of the 3 subtests of the WNV (i.e. matrices, recognition, and coding for patients aged <8 years and matrices, spatial span, and coding for patients aged 8 to 21 years). The composite WNV score has no range.
Time Frame: Baseline, Week 18
Population: The safety Set comprised all patients who received at least one dose of study treatment and had at least one post-baseline safety assessment in the Core phase (where the statement that a patient had no AE constitutes a safety assessment.
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo | Everolimus Long Term Evaluation (LTE)
Number analyzed (Participants) | 89 | 94 | 85 | 0
scores on a scale
  Baseline: number analyzed (Participants) | 63 | 63 | 52 | 0
  Baseline | -0.48 [-2.3 to 8.1] | -0.69 [-2.3 to 9.6] | -1.11 [-2.3 to 8.3] |
  End of Core Phase: number analyzed (Participants) | 60 | 63 | 48 | 0
  End of Core Phase | -0.04 [-2.3 to 8.1] | -0.89 [-2.3 to 7.5] | -0.51 [-2.3 to 10.1] |
  Change from Baseline: number analyzed (Participants) | 58 | 59 | 46 | 0
  Change from Baseline | 0.00 [-2.5 to 1.6] | 0.00 [-10.0 to 2.1] | 0.00 [-3.3 to 1.7] |

14. Secondary Outcome: Long Term Evaluation: Effect of Everolimus Over Time in the Overall Wechsler Nonverbal Composite Score
Description: as for outcome 13
Time Frame: Baseline, Weeks 18, 42, 66 and 90
Population: as for outcome 12
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo | Everolimus Long Term Evaluation (LTE)
Number analyzed (Participants) | 0 | 0 | 0 | 265
scores on a scale
  Baseline: number analyzed (Participants) | 0 | 0 | 0 | 151
  Baseline |  |  |  | -0.53 [-2.3 to 10.1]
  Week 18: number analyzed (Participants) | 0 | 0 | 0 | 160
  Week 18 |  |  |  | -0.44 [-2.3 to 9.5]
  Week 42: number analyzed (Participants) | 0 | 0 | 0 | 139
  Week 42 |  |  |  | -0.36 [-2.3 to 10.8]
  Week 66: number analyzed (Participants) | 0 | 0 | 0 | 104
  Week 66 |  |  |  | 0.13 [-2.3 to 9.1]
  Week 90: number analyzed (Participants) | 0 | 0 | 0 | 82
  Week 90 |  |  |  | -0.06 [-2.3 to 9.0]

15. Secondary Outcome: Core Phase: Response Rate in Seizure Frequency by Time Normalized Minimum Concentration
Description: Comparison of response rate in seizure frequency for 5 categories of time-normalized minimum concentration (Cmin, TN) (< 3 ng/mL; 3-7 ng/mL; >7-<9 ng/mL; 9-15 ng/mL; >15 ng/mL). Response rate is the percentage of patients with ≥ 50% reduction from baseline in average weekly partial-onset seizure frequency during the maintenance period of the Core phase.
Time Frame: Baseline (8-week period before randomization), Week 7 to 18 (12-week maintenance period of the core phase)
Population: Confirmed PK Sample Set from all everolimus-treated patients in the Safety Set was defined as: Cmin collected prior to dose administration on the same treatment day and 20-28 hours after the previous dose, at steady state, and with no evidence of vomiting within 4 hours of the previous dose.
Measure: Median (95% Confidence Interval); unit: Percentage of responders
Groups:
- <3 ng/mL: Observed TN-Cmin concentration during the maintenance of the core phase: <3 ng/mL
- 3-7 ng/mL: Observed TN-Cmin concentration during the maintenance of the core phase:3 - 7 ng/mL
- >7-<9 ng/mL: Observed TN-Cmin concentration during the maintenance of the core phase: >7 - <9 ng/mL
- 9-15 ng/mL: Observed TN-Cmin concentration during the maintenance of the core phase: 9 - 15 ng/mL
- >15 ng/mL: Observed TN-Cmin concentration during the maintenance of the core phase: >15 ng/mL
Arm/Group | <3 ng/mL | 3-7 ng/mL | >7-<9 ng/mL | 9-15 ng/mL | >15 ng/mL
Number analyzed (Participants) | 14 | 147 | 52 | 30 | 2
Percentage of responders | 14.3 [1.8 to 42.8] | 29.9 [22.7 to 38.0] | 44.2 [30.5 to 58.7] | 50.0 [31.3 to 68.7] | 50.0 [1.3 to 98.7]

16. Secondary Outcome: Core Phase: Median Percentage Change From Baseline in Seizure Frequency by Time Normalized Minimum Concentration
Description: Percentage change from baseline in average weekly seizure frequency during the maintenance period of the Core phase is calculated as follow: (SFcfb) = 100 × (SFB - SFM) ÷ SFB where SFB is the average weekly seizure frequency in the Baseline phase and SFM is the average weekly seizure frequency in the maintenance period of the Core phase. A positive percentage change from baseline (SFcfb) means a reduction in seizure frequency whereas a negative percentage change from baseline (SFcfb) means an increase in seizure frequency.
Time Frame: Baseline (8-week period before randomization), Week 7 to 18 (12-week maintenance period of the core phase)
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: Percentage change
Arm/Group | <3 ng/mL | 3-7 ng/mL | >7-<9 ng/mL | 9-15 ng/mL | >15 ng/mL
Number analyzed (Participants) | 14 | 147 | 52 | 30 | 2
Percentage change | 20.55 [-8.45 to 35.39] | 35.56 [24.43 to 41.88] | 39.72 [28.02 to 62.79] | 47.69 [36.46 to 66.32] | 61.56 [42.73 to 80.38]

17. Secondary Outcome: Long Term Evaluation: Relationship Between Seizure Frequency and Time-normalized Everolimus Concentration at Trough (Cmin,TN) - Repeated Measures Analysis
Description: A repeated measures analysis considering fixed 2-week intervals and including the level of exposure (time-normalized Cmin values), the time on-treatment and the seizure frequency at baseline quantified the estimated percentage change over 2 weeks in seizure frequency associated with a double exposure to everolimus, 15 days more on treatment and half the seizure frequency at baseline. A positive percentage change means a reduction in seizure frequency whereas a negative percentage change means an increase in seizure frequency.
Time Frame: During everolimus treatment from start of everolimus up to the end of the extension phase, an average of 1.7 year
Population: Confirmed PK Sample Set from all everolimus-treated patients in the Longer-term Evaluation (LTE) Safety Set, was defined as follows: Cmin collected prior to dose administration on the same treatment day and 20-28 hours after the previous dose, at steady state, and with no evidence of vomiting within 4 hours of the previous dose
Measure: Mean (95% Confidence Interval); unit: % change over 2-wk in seizures freq.
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo | Everolimus Long Term Evaluation (LTE)
Number analyzed (Participants) | 0 | 0 | 0 | 358
% change over 2-wk in seizures freq.
  By doubling the time-normalized Cmin (log scale) |  |  |  | 8.93 [6.87 to 10.95]
  By reporting half the seizure freq. at baseline |  |  |  | 48.82 [46.37 to 51.15]
  By adding 12 weeks on treatmen |  |  |  | 6.42 [4.53 to 8.27]

18. Secondary Outcome: Core Phase: Impact of Everolimus on Anti-epileptic Drugs (AEDs) Concentrations
Description: Impact of everolimus on AED concentrations at trough. Pre-dose plasma samples to measure AED concentrations were measured at at Visits 1 (Screening), 2 (Baseline), 3, and 5. Effects of everolimus on the exposure of antiepileptic drugs was assessed by comparing the anti-epileptic drug concentrations at Visits 1 and 2 (AEDs alone) and at Visits 3 and 5 (AEDs plus everolimus).
Time Frame: Baseline, Weeks 1 & 3
Population: Confirmed PK Sample Set from all everolimus-treated patients in the Safety Set and Long-term Evaluation (LTE) Safety Set was defined as: Cmin collected prior to dose administration on the same treatment day and 20-28 hours after the previous dose, at steady state, and with no evidence of vomiting within 4 hours of the previous dose.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Valporic Acid; Carbamazepine; Clobazam; N-desmethylclobazam; Topiramate; TRI477; TRI476; Clonazepam; Zonisamide; Phenobarbital; Phenytoin: Antiepileptic drug
Arm/Group | Valporic Acid | Carbamazepine | Clobazam | N-desmethylclobazam | Topiramate | TRI477 | TRI476 | Clonazepam | Zonisamide | Phenobarbital | Phenytoin
Number analyzed (Participants) | 86 | 34 | 37 | 37 | 34 | 31 | 31 | 17 | 12 | 11 | 7
ng/mL | 0.962 [0.913 to 1.014] | 1.108 [1.016 to 1.208] | 1.093 [1.037 to 1.153] | 1.071 [1.017 to 1.127] | 0.983 [0.872 to 1.108] | 1.086 [0.913 to 1.291] | 1.194 [0.936 to 1.523] | 1.065 [0.974 to 1.163] | 1.028 [0.971 to 1.089] | 0.957 [0.886 to 1.034] | 1.020 [0.874 to 1.190]

19. Secondary Outcome: Long Term Evaluation: Percentage Change From Start of Everolimus in Seizure Frequency by Time Window
Description: Percentage change from start of everolimus in average weekly seizure frequency (SFcfe) = 100 × (SFe - SFtw) ÷ SFe where:
  SFe is the average weekly seizure frequency in the 8-week period before start of everolimus SFtw is the average weekly seizure frequency in a 12-week time window A positive percentage change from start of everolimus (SFcfe) means a reduction in seizure frequency whereas a negative percentage change from start of everolimus (SFcfe) means an increase in seizure frequency.
Time Frame: Baseline (8-week period before start of everolimus), Week 7 to 18, Week 19 to 30, and 12 weeks thereafter up to Week 102
Population: The LTE Efficacy Set included 361 patients who received at least one dose of everolimus in Core and Extension phase and had at least one valid postbaseline efficacy evaluation.
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo | Everolimus Long Term Evaluation (LTE)
Number analyzed (Participants) | 0 | 0 | 0 | 361
Percent change
  Week 18: number analyzed (Participants) | 0 | 0 | 0 | 352
  Week 18 |  |  |  | 31.65 [28.51 to 36.09]
  Week 30: number analyzed (Participants) | 0 | 0 | 0 | 335
  Week 30 |  |  |  | 35.74 [29.37 to 39.06]
  Week 42: number analyzed (Participants) | 0 | 0 | 0 | 320
  Week 42 |  |  |  | 42.86 [34.44 to 48.15]
  Week 54: number analyzed (Participants) | 0 | 0 | 0 | 299
  Week 54 |  |  |  | 46.05 [39.93 to 53.61]
  Week 66: number analyzed (Participants) | 0 | 0 | 0 | 282
  Week 66 |  |  |  | 49.07 [38.26 to 55.56]
  Week 78: number analyzed (Participants) | 0 | 0 | 0 | 252
  Week 78 |  |  |  | 51.69 [43.88 to 61.58]
  Week 90: number analyzed (Participants) | 0 | 0 | 0 | 222
  Week 90 |  |  |  | 57.33 [47.37 to 67.01]
  Week 102: number analyzed (Participants) | 0 | 0 | 0 | 191
  Week 102 |  |  |  | 59.69 [52.13 to 70.94]

20. Secondary Outcome: Seizure Free Rates by Time Window
Description: Percentage of seizure-free participants for each 12-week time window.
Time Frame: Weeks 18, 30, 42, 54, 66, 78, 90 & 102
Population: The LTE Efficacy Set included 361 patients who received at least one dose of everolimus in Core and Extension phase and had at least one valid post baseline efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: Percentage of seizure-free participants
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo | Everolimus Long Term Evaluation (LTE)
Number analyzed (Participants) | 0 | 0 | 0 | 361
Percentage of seizure-free participants
  Week 18: number analyzed (Participants) | 0 | 0 | 0 | 352
  Week 18 |  |  |  | 3.98 [2.2 to 6.6]
  Week 30: number analyzed (Participants) | 0 | 0 | 0 | 335
  Week 30 |  |  |  | 6.87 [4.4 to 10.1]
  Week 42: number analyzed (Participants) | 0 | 0 | 0 | 320
  Week 42 |  |  |  | 8.44 [5.6 to 12.0]
  Week 54: number analyzed (Participants) | 0 | 0 | 0 | 299
  Week 54 |  |  |  | 8.70 [5.8 to 12.5]
  Week 66: number analyzed (Participants) | 0 | 0 | 0 | 282
  Week 66 |  |  |  | 10.99 [7.6 to 15.2]
  Week 78: number analyzed (Participants) | 0 | 0 | 0 | 252
  Week 78 |  |  |  | 13.49 [9.5 to 18.3]
  Week 90: number analyzed (Participants) | 0 | 0 | 0 | 222
  Week 90 |  |  |  | 14.86 [10.5 to 20.2]
  Week 102: number analyzed (Participants) | 0 | 0 | 0 | 191
  Week 102 |  |  |  | 15.18 [10.4 to 21.1]

21. Secondary Outcome: Core Phase: Incidence of Suicide Attempt, Suicidal Ideation or Behavior During Core Phase Per Columbia Suicide Severity Rating Scale (C-SSRS) Outcomes
Description: Comparison of suicidality using the C-SSRS in the everolimus low-trough treatment arm (3-7 ng/mL), high-trough treatment arm (9-15 ng/mL) and placebo arm. The Columbia-Suicide Severity Rating Scale (C-SSRS) is a questionnaire used for suicide assessment developed by multiple institutions, including Columbia University, with NIMH support. The scale is evidence-supported and is part of a national and international public health initiative involving the assessment of suicidality. There are different scoring systems depending on the population. The important elements to note are that the higher the scores on the individual items and the more "yes" items, the higher the suicide risk.
Time Frame: Baseline, Week 18
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo
Number analyzed (Participants) | 117 | 130 | 119
Participants
  Completed suicide | 0 | 0 | 0
  Suicide attempt | 1 | 0 | 0
  Prep actions toward imminent suicidal behavior | 2 | 0 | 0
  Suicidal ideation | 3 | 1 | 0
  Self-injurious behavior without suicide intent | 0 | 0 | 0

22. Secondary Outcome: Long Term Evaluation: Incidence of Suicide Attempt, Suicidal Ideation or Behavior During Core Phase Per Columbia Suicide Severity Rating Scale (C-SSRS) Outcomes
Description: The C-SSRS was completed at each visit. The table below presents the number of patients who reported at least one completed suicide, one suicide attempt, one preparatory action toward imminent suicidal behavior, one suicidal ideation and one self-injurious behavior without suicidal intent at any time point after starting everolimus.
Time Frame: During everolimus treatment from start of everolimus up to permanent discontinuation of everolimus, an average of 2.3 years
Population: The LTE Efficacy Set included 361 patients who received at least one dose of everolimus in Core and Extension phase and had at least one valid post-baseline efficacy evaluation.
Measure: Number; unit: Participants
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Placebo | Everolimus Long Term Evaluation (LTE)
Number analyzed (Participants) | 0 | 0 | 0 | 361
Participants
  Completed suicide |  |  |  | 0
  Suicidal attempt |  |  |  | 1
  Prep. actions toward imminent suicidal behavior |  |  |  | 2
  Suicidal ideation |  |  |  | 7
  Self-injurious behavior without suicide intent |  |  |  | 1

ADVERSE EVENTS:
Time Frame: Adverse Events were collected during everolimus treatment from start of everolimus up to permanent discontinuation of everolimus, an average of 2.3 years
Description: The summary tables below include all adverse events starting or worsening on or after the first dose of everolimus, and starting no later than 30 days after the date of last dose of everolimus. Adverse events starting during the placebo period were not counted.
Groups:
- Everolimus Start Ext: Participants who received placebo dispersible tablets for oral suspension at study start and switched to everolimus in Extension.
- Everolimus All: Participants who were treated with everolimus either in the Core or Extension phases of the study and were evaluated for longer term safety and efficacy.
Arm/Group | Everolimus LT Target of 3 to 7 ng/mL | Everolimus HT Target of 9 to 15 ng/mL | Everolimus Start Ext | Everolimus All
All-Cause Mortality (participants affected / at risk) | 1/117 | 2/130 | 1/114 | 4/361
Serious Adverse Events (participants affected / at risk) | 50/117 | 49/130 | 38/114 | 137/361
Other Adverse Events (participants affected / at risk) | 110/117 | 126/130 | 109/114 | 345/361
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus LT Target of 3 to 7 ng/mL (N=117) | Everolimus HT Target of 9 to 15 ng/mL (N=130) | Everolimus Start Ext (N=114) | Everolimus All (N=361)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Blepharitis (Eye disorders) | 1 | 0 | 0 | 1
Meibomianitis (Eye disorders) | 1 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 1
Retinopathy proliferative (Eye disorders) | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 0 | 5
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastric ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 3 | 0 | 1 | 4
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 1 | 4
Swollen tongue (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 4
Asthenia (General disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 0 | 2
Pyrexia (General disorders) | 5 | 4 | 2 | 11
Sudden unexplained death in epilepsy (General disorders) | 0 | 2 | 0 | 2
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 1 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 3 | 2 | 6
Campylobacter colitis (Infections and infestations) | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 2 | 3
Corona virus infection (Infections and infestations) | 0 | 1 | 0 | 1
Croup infectious (Infections and infestations) | 1 | 2 | 0 | 3
Dacryocanaliculitis (Infections and infestations) | 1 | 0 | 0 | 1
Ear infection (Infections and infestations) | 1 | 0 | 1 | 2
Febrile infection (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 5 | 5 | 4 | 14
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1 | 2
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 0 | 1 | 1
Herpangina (Infections and infestations) | 1 | 1 | 0 | 2
Influenza (Infections and infestations) | 3 | 1 | 2 | 6
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 2
Lung infection (Infections and infestations) | 1 | 0 | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 0 | 1 | 1
Meningitis (Infections and infestations) | 0 | 0 | 1 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 2 | 0 | 2
Otitis media (Infections and infestations) | 0 | 0 | 1 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 1 | 1 | 4
Pharyngitis streptococcal (Infections and infestations) | 0 | 2 | 0 | 2
Pneumonia (Infections and infestations) | 16 | 13 | 9 | 38
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 1 | 2
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 2 | 0 | 1 | 3
Pneumonia viral (Infections and infestations) | 0 | 1 | 2 | 3
Pseudocroup (Infections and infestations) | 1 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 2 | 2 | 0 | 4
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Rotavirus infection (Infections and infestations) | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 1 | 0 | 2
Septic shock (Infections and infestations) | 0 | 1 | 1 | 2
Sinusitis (Infections and infestations) | 1 | 1 | 1 | 3
Skin infection (Infections and infestations) | 0 | 1 | 1 | 2
Tonsillitis (Infections and infestations) | 0 | 2 | 3 | 5
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 0 | 0 | 3
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 1
Varicella (Infections and infestations) | 1 | 0 | 1 | 2
Viraemia (Infections and infestations) | 0 | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 0 | 3 | 3
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 3
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Tongue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 1
Urine output decreased (Investigations) | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Feeding intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 2 | 3
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Dyskinesia (Nervous system disorders) | 1 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 2 | 0 | 0 | 2
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 1 | 2
Headache (Nervous system disorders) | 0 | 2 | 0 | 2
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 1
Moyamoya disease (Nervous system disorders) | 0 | 1 | 0 | 1
Seizure (Nervous system disorders) | 7 | 7 | 4 | 18
Seizure cluster (Nervous system disorders) | 1 | 0 | 0 | 1
Status epilepticus (Nervous system disorders) | 7 | 6 | 2 | 15
Stupor (Nervous system disorders) | 1 | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0 | 1
Affect lability (Psychiatric disorders) | 0 | 0 | 1 | 1
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 1
Mood altered (Psychiatric disorders) | 1 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1
Post streptococcal glomerulonephritis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Sexual abuse (Social circumstances) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus LT Target of 3 to 7 ng/mL (N=117) | Everolimus HT Target of 9 to 15 ng/mL (N=130) | Everolimus Start Ext (N=114) | Everolimus All (N=361)
Anaemia (Blood and lymphatic system disorders) | 10 | 7 | 4 | 21
Neutropenia (Blood and lymphatic system disorders) | 4 | 9 | 1 | 14
Abdominal pain (Gastrointestinal disorders) | 10 | 4 | 5 | 19
Abdominal pain upper (Gastrointestinal disorders) | 7 | 10 | 5 | 22
Aphthous ulcer (Gastrointestinal disorders) | 11 | 23 | 10 | 44
Constipation (Gastrointestinal disorders) | 9 | 12 | 7 | 28
Dental caries (Gastrointestinal disorders) | 6 | 2 | 3 | 11
Diarrhoea (Gastrointestinal disorders) | 45 | 42 | 30 | 117
Mouth ulceration (Gastrointestinal disorders) | 36 | 44 | 22 | 102
Nausea (Gastrointestinal disorders) | 6 | 7 | 3 | 16
Stomatitis (Gastrointestinal disorders) | 41 | 48 | 41 | 130
Vomiting (Gastrointestinal disorders) | 28 | 35 | 16 | 79
Fatigue (General disorders) | 8 | 11 | 5 | 24
Pyrexia (General disorders) | 47 | 56 | 31 | 134
Bronchitis (Infections and infestations) | 11 | 17 | 8 | 36
Conjunctivitis (Infections and infestations) | 11 | 8 | 6 | 25
Ear infection (Infections and infestations) | 11 | 19 | 3 | 33
Gastroenteritis (Infections and infestations) | 13 | 15 | 7 | 35
Gingivitis (Infections and infestations) | 9 | 4 | 0 | 13
Hordeolum (Infections and infestations) | 6 | 5 | 4 | 15
Influenza (Infections and infestations) | 16 | 18 | 9 | 43
Lower respiratory tract infection (Infections and infestations) | 7 | 1 | 2 | 10
Nasopharyngitis (Infections and infestations) | 33 | 35 | 26 | 94
Pharyngitis (Infections and infestations) | 11 | 18 | 8 | 37
Respiratory tract infection (Infections and infestations) | 3 | 0 | 6 | 9
Rhinitis (Infections and infestations) | 9 | 9 | 5 | 23
Sinusitis (Infections and infestations) | 3 | 15 | 8 | 26
Tonsillitis (Infections and infestations) | 11 | 9 | 4 | 24
Upper respiratory tract infection (Infections and infestations) | 32 | 42 | 22 | 96
Urinary tract infection (Infections and infestations) | 12 | 10 | 6 | 28
Viral infection (Infections and infestations) | 9 | 7 | 2 | 18
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 7 | 1 | 10
Contusion (Injury, poisoning and procedural complications) | 5 | 8 | 3 | 16
Fall (Injury, poisoning and procedural complications) | 15 | 10 | 8 | 33
Laceration (Injury, poisoning and procedural complications) | 3 | 4 | 6 | 13
Skin abrasion (Injury, poisoning and procedural complications) | 6 | 5 | 2 | 13
Blood cholesterol increased (Investigations) | 14 | 20 | 17 | 51
Blood triglycerides increased (Investigations) | 5 | 10 | 6 | 21
Low density lipoprotein increased (Investigations) | 6 | 8 | 3 | 17
Weight decreased (Investigations) | 10 | 7 | 8 | 25
Decreased appetite (Metabolism and nutrition disorders) | 13 | 20 | 6 | 39
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 | 9 | 2 | 15
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 9 | 12 | 6 | 27
Headache (Nervous system disorders) | 19 | 19 | 10 | 48
Somnolence (Nervous system disorders) | 8 | 9 | 4 | 21
Aggression (Psychiatric disorders) | 5 | 8 | 1 | 14
Agitation (Psychiatric disorders) | 7 | 1 | 2 | 10
Insomnia (Psychiatric disorders) | 8 | 8 | 2 | 18
Irritability (Psychiatric disorders) | 5 | 4 | 7 | 16
Menstruation irregular (Reproductive system and breast disorders) | 1 | 7 | 3 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 33 | 15 | 77
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 12 | 3 | 19
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 1 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 10 | 5 | 20
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10 | 9 | 3 | 22
Acne (Skin and subcutaneous tissue disorders) | 6 | 14 | 6 | 26
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 8 | 2 | 14
Dermatitis (Skin and subcutaneous tissue disorders) | 7 | 2 | 2 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 3 | 2 | 11
Rash (Skin and subcutaneous tissue disorders) | 14 | 21 | 13 | 48
Hypertension (Vascular disorders) | 6 | 7 | 6 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2016-03-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT01713946/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT01713946/SAP_001.pdf